CLINICAL TRIAL: NCT01980784
Title: Posttraumatic Changes in Energy Expenditure and Body Composition in Patients With Acute Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Principal Investigator, Intensivmedizin SPZ, Dr. Peter Felleiter, Swiss Paraplegic Research, Nottwil
Other Study IDs: 2012-08
Record Dates: First submitted 2013-10-17; First posted 2013-11-11 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Severe trauma induces massive metabolic changes that are characterized by hypermetabolism with increased energy expenditure and catabolism. Early enteral and, if necessary, parenteral feeding is a major focus of modern intensive care medicine.

After acute spinal cord injury, denervation of skeletal muscle leads to a massive loss of muscle mass in the area below the level of injury. This dramatic muscle atrophy again leads to a decrease in energy expenditure. Whereas other survivors of severe trauma typically regain muscle mass during rehabilitation, spinal cord injury patients typically continue to lose muscle mass over time, which also leads to changes in body composition. The time course of these changes is not known. Continuing nutrition without adaption to the reduced energy expenditure leads to weight gain and adiposity, exposing many chronic spinal cord injury patients to the known unfavorable metabolic consequences. Knowledge of the time course of these changes would help to provide adequate caloric intake to the patients and improve our ability for nutrition counseling.

The investigators plan a prospective clinical trial in 25 acute spinal cord injury patients to determine the changes in energy expenditure and body composition. Major inclusion criteria are acute traumatic spinal cord injury, age 18-70, neurological level above L1, AIS (American Spinal Injury Association Impairment Scale) A, B or C.

Measurements of energy expenditure, body composition and nutritional markers in venous blood are scheduled 2, 6, 10 and 14 weeks after spinal cord injury and at the end of rehabilitation (at the latest after 26 weeks).

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for acute treatment and rehabilitation after traumatic spinal cord injury
* no longer then two weeks after onset of spinal cord injury
* age 18 - 70 years
* body mass index 18-30
* neurological level C4 to Th12
* American Spinal Injury Association Impairment Scale (AIS) A, B or C

Exclusion Criteria:

* complications during acute treatment, which make study participation impossible or would endanger the recovery of the patient
* pre-existing diabetes mellitus type 1 and 2
* pre-existing hypercholesterolemia
* untreated hypothyroidism or hyperthyroidism
* invasive mechanical ventilation
* cardiac pacemaker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of a spinal cord injury rehabilitation centre
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes in energy expenditure | 2, 6, 10, 14 and 26 weeks after spinal cord injury
  Resting energy expenditure [kcal/day] measured by indirect calorimetry.

SECONDARY OUTCOMES:
Changes in body composition | 2, 6, 10, 14 and 26 weeks after spinal cord injury
  Body composition measured by bioelectric impedance analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre Nottwil, Nottwil, Canton of Lucerne, Switzerland